CLINICAL TRIAL: NCT05391009
Title: Comparison of PNF and Task Related Techniques Along With Tens on Upper Limb Function Among Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/513
Record Dates: First submitted 2022-05-09; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF GROUP (Experimental): PNF exercise twice daily five days per week for 8 weeks. D1 and D2 flexion and extension pattern for upper limb. In D1 Flexion-adduction -external rotation d1, extension -abduction-internal rotation and in D2 flexion-abduction-external rotation, extension-adduction-internal rotation
  Interventions: Diagnostic Test: PNF
- TRT GROUP (Experimental): The duration of a TRT session Will be 60 min. Each session started with warm-up exercises for 10 min followed by 50 min of TRT. Each task will be repeated approximately 10 to 20 times, for 1 to 5 sets, or alternatively for 2 to 5 min. A 2 min rest period after every 15 min of practice will be allowed. Before commencing the exercise session, tasks will be demonstrated to each patient using the non-affected UE.
  Interventions: Diagnostic Test: TRT

INTERVENTIONS:
Diagnostic Test: PNF — PNF exercise twice daily five days per week for 8 weeks. D1 and D2 flexion and extension pattern for upper limb. In D1 Flexion-adduction -external rotation d1, extension -abduction-internal rotation and in D2 flexion-abduction-external rotation, extension-adduction-internal rotation
  Arms: PNF GROUP
Diagnostic Test: TRT — The duration of a TRT session Will be 60 min. Each session started with warm-up exercises for 10 min followed by 50 min of TRT. Each task will be repeated approximately 10 to 20 times, for 1 to 5 sets, or alternatively for 2 to 5 min. A 2 min rest period after every 15 min of practice will be allowed. Before commencing the exercise session, tasks will be demonstrated to each patient using the non-affected UE.
  Arms: TRT GROUP

SUMMARY:
Comparison of PNF and Task Related Techniques Along with Tens on Upper Limb Function Among Stroke Patients

DETAILED DESCRIPTION:
The objective of this study is to determine the comparison of PNF and TRT along with TENs on upper limb function recovery among stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Duration of illness before participation in the study ranged from six to eighteen months' post stroke.
* Patients who diagnosed with ischemic stroke stage 2 and 3
* Patients' age ranged from 50-70 years (male/female)
* Patients with sufficient cognitive abilities that enables them to understand and follow instructions (mini mental scale)

Exclusion Criteria:

* Patients with communication problems
* Patients with a history of previous stroke or other neurological diseases or disorders
* Patients with inflammation, old fracture or prosthesis in the affected limb, neurological diseases that affect upper limb function other than stroke (e.g.: Multiple sclerosis, Peripheral neuropathy, Parkinsonism .... etc.), infection or dermatological conditions on acupuncture sites, musculoskeletal disorders such as severe arthritis, cardiovascular problems (unstable angina, recent myocardial infarction within the last three months, congestive heart failure, significant heart valve dysfunction, arrhythmia, implanted pacemaker or unstable hypertension) or pulmonary disorders, visual and auditory problems and patients with cognitive impairment.
* Any Contra indications for TENS, Other neurological & orthopedic conditions affecting upper limb, Patient with subluxed shoulder, Patient with shoulder hand syndrome.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Task Related Techniques Along With Tens on Upper Limb Function Among Stroke Patients | 6 Months
  The duration of a TRT session Will be 60 min. Each session started with warm-up exercises for 10 min followed by 50 min of TRT. Modified ashworth scale (mas) Box and block test

SECONDARY OUTCOMES:
PNF Techniques Along With Tens on Upper Limb Function Among Stroke Patients | 6 Months
  PNF exercise twice daily five days per week for 8 weeks. D1 and D2 flexion and extension pattern for upper limb. Mini Mental Scale

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital, Al Shafi hospital, CH. Muhammad Akram Hospital Hameed Latif Hospital., Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No